CLINICAL TRIAL: NCT01344967
Title: Suppression of Bone Turnover Following Treatment With Zoledronic Acid in Patients With Metastatic Breast Cancer: Duration of Effect
Acronym: SuBDuE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHN-080520C
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Metastatic Breast Cancer With Bone Involvement
MeSH Terms: interventions — Zoledronic Acid

ARMS (1):
- Zometa, Bone Suppression, Active Ingredient (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic Acid at a dose of 4mg will be administered by intravenous infusion over 15 minutes in at least 100mls of saline
  Other Names: Control No. 110322

SUMMARY:
Bone is the most common site of spread of breast cancer and bone metastases will occur in roughly 70% of women with advanced disease. These patients are at risk of developing bone complications that cause significant impact on both patient morbidity and mortality. Close to two-thirds of women with bone metastases will go on to develop at least one of these complications, termed a skeletal related event (SRE), defined as 1) pathological fractures, 2) pain requiring radiation or surgical intervention, 3)spinal cord compression, and 4) hypercalcemia. In addition to SREs, most breast cancer patients with bone metastases have some degree of pain associated with their disease. Understandably these factors negatively impact their quality of life. Furthermore, the development of an SRE in this population has been shown to be associated with shorter overall survival. Prevention or delay in onset of these complications is therefore an important therapeutic goal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed breast cancer.
2. Radiological or pathological evidence of bone metastases. (positive bone scan, MRI, or CT or pathological fracture, or pathological sample from bone biopsy showing evidence of metastatic breast cancer).
3. Patient has not yet started on BP therapy for metastatic breast cancer to bone.
4. Renal (serum creatinine, BUN), hepatic (AST, ALT, Bilirubin) function within the institutional normal range as assessed within 1 month of study entry.
5. Age >/= 18 years.
6. Karnofsky performance status ≥ 50.
7. Life expectancy > 6 months.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients may receive any chemotherapy, biological or endocrine treatment considered appropriate by the treating physician. This can be changed during the course of the study as clinically indicated.
10. Patients may be on another clinical trial, if allowed by the Trial Steering Committee for that trial.
11. Patients are willing to take calcium and vitamin D supplements as recommended, while on study.

Exclusion Criteria:

1. Hypersensitivity or known allergy to bisphosphonates.
2. Patient currently taking Bisphosphonate therapy for metastatic breast cancer to bone (Clodronate, Pamidronate, Zoledronic Acid, Ibandronate, Calcitonin). Bisphosphonates for the treatment of other bone disease (osteoporosis, osteopenia, Paget's disease, etc) but not Zoledronic Acid, are permitted.
3. Acute or chronic renal insufficiency.
4. Hypocalcemia as defined by serum calcium less than institutional normal range.
5. Evidence of infection/abscess on dental exam or recent dental extraction (within last 4 weeks), or presence of osteonecrosis of the jaw.
6. Acute pathological fracture, spinal cord compression, or hypercalcemia requiring urgent treatment (patient may enter study after acute issues are resolved).
7. Patients with baseline hypocalcemia.
8. Patients who have received ZA for prevention of breast cancer treatment-induced osteopenia or osteoporosis within the last 1 year.
9. History and/or electrocardiographic evidence of atrial fibrillation.
10. Pregnancy or lactation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to estimate the proportion of patients with suppression of bone turnover at 12 weeks after administration of a single dose of Zoledronic Acid | Baseline to Twelve weeks

SECONDARY OUTCOMES:
To estimate the distribution of duration of suppression of bone turnover up to 12 weeks after administration of Zoledronic Acid | Baseline to Twelve weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada